CLINICAL TRIAL: NCT06381297
Title: The Effect Of Medial Olivocochlear Efferents On Speech Discrimination In Noise In Multiple Sclerosis.
Brief Title: Speech in Noise Discrimination Skills in Multiple Sclerosis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asuman Kucukoner (Other)
Responsible Party: Sponsor-Investigator, Asuman Kucukoner, Lecturer, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: OndokusMU; Ondokuz Mayıs University (Registry Identifier: Clinical research ethics committee)
Record Dates: First submitted 2024-04-01; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis-Relapsing-Remitting
Keywords: Multıple sclerosis,; Auditory efferent system; Contralateral supression; speech in noise discrimination
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Hearing Tests

STUDY DESIGN:
Intervention Model Description: Multiple sclerosis patient group and healthy control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS group (Active Comparator): Study group (MS patients)
  Interventions: Diagnostic Test: Hearing test; Diagnostic Test: Speech in noise discrimination test; Diagnostic Test: Montreal Cognitive Assessment Scale; Diagnostic Test: Symbol Number Modalities Test (SDMT)
- Control group (Placebo Comparator): Control group ( Healty individuals)
  Interventions: Diagnostic Test: Hearing test; Diagnostic Test: Speech in noise discrimination test; Diagnostic Test: Montreal Cognitive Assessment Scale; Diagnostic Test: Symbol Number Modalities Test (SDMT)

INTERVENTIONS:
Diagnostic Test: Hearing test — Hearing and speech tests of MS group and control group in the presence and absence of noise will be evaluated. Suppression test will be performed with OAE test in the presence and absence of noise.
  Other Names: Contralateral supression test
Diagnostic Test: Speech in noise discrimination test — Speech discrimination in noise (SDN) test will be performed in a quiet room in accordance with the Industrial Acoustic Company (IAC) standard using the Grason-Stadler GSI 61 Clinical Audiometer. After pure tone audiometry and speech tests, the GKAE test will be performed. The speech in noise discrimination test will be performed with a signal-to-noise (S/N) ratio of +10 dB. A word list at 50 dB SL will be presented to the tested ear using live sound, while simultaneously white noise at 40 dB SL will be presented to the test ear (Beattie et al. 1997). This will be done for both ears. The speech in noise discrimination test scores will be calculated as percentages (%) for both ears.
Diagnostic Test: Montreal Cognitive Assessment Scale — Translated into Turkish as the Montreal Cognitive Assessment Scale and abbreviated as MOBID, MOCA assesses attention, executive/managerial functions, memory, visual-spatial skills, language, abstract thinking and arithmetic. It is easy and practical to apply. The score that can be obtained varies between 0-30. The cut-off point for cognitive impairment is 21. Patients who perform below 21 points are considered to have cognitive impairment. Although it is not a battery used in the MS patient group, a study conducted on 39 MS patients and 20 healthy people showed that it can be used safely for screening purposes in patients with MS (Aksoy et al., 2013; Nasreddine et al., 2005; Selekler & Cangoz, 2009).
Diagnostic Test: Symbol Number Modalities Test (SDMT) — Attention, visuospatial information processing speed and working memory are assessed. It is one of the subtests of the Short Repeatable Neuropsychological Battery developed to assess cognitive functions in MS (Smith, 1973).

SUMMARY:
The aim of this clinical trial was to determine the effect of multiple sclerosis on speech reception and discrimination in noise and to compare the effects on the medial olivocochlear reflex, which is thought to affect speech intelligibility in noise, with a control group.

The main questions it aims to answer are:

Does MS disease affect the ability to discriminate speech in noise? Does MS affect contralateral suppression results assessing medial olivocochlear function? Is there a correlation between the ability to discriminate speech in noise and contralateral suppression skills of MS patients? Data from MS patients and healthy participants will be compared. Thirty relapsing remitting MS patients and 30 healthy participants admitted to the clinic will be evaluated.

DETAILED DESCRIPTION:
The second aim was to evaluate the relationship between speech comprehension and discrimination skills in noise and cognitive function and to compare them with the control group.

Inclusion Criteria for the Study Group

1. Being diagnosed with MS (Primary Progressive, Secondary Progressive, Relapsing Remittting) - exclusion criteria for the control group
2. Being between 18-50 years old
3. Volunteering
4. Co-operation with the scales and tests to be applied
5. Normal ENT otoscopic (external and middle ear) examination findings
6. Having a normal (type A) tympanogram with a peak value of ± 50 daPa on acoustic impedancemetry examination
7. Pure voice average within normal limits (Clark, 1981).
8. Speech scores within normal limits (Jerger & Hayes, 1977).
9. No other neurological, psychiatric, metabolic diseases other than MS
10. No history of noise exposure and ototoxic drug use Exclusion Criteria for Volunteers

1) Not diagnosed with MS (Primary Progressive, Secondary Progressive, Relapsing Remittting) - inclusion criteria for the control group 2) Being younger than 18 years old and older than 50 years old 3) Not wanting to participate in the study or giving up participation 4) Inability to cooperate with the scales and tests to be applied 5) Detection of pathology in ENT otoscopic (external and middle ear) examination findings 6) Obtaining Type B and Type C tympanograms 7) Hearing loss 8) Speech scores are not normal 9) Having any neurological, psychiatric, metabolic disease - MS diagnosis is the inclusion criterion for the study group 10) History of noise exposure and ototoxic drug use The primary endpoint of the study will be to evaluate whether there is a relationship between the MOC reflex and the thresholds for speech reception and discrimination in noise in individuals diagnosed with MS.

It will be evaluated whether cognitive function differences in individuals diagnosed with MS show differences in speech in noise and discrimination thresholds.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Relapsing-remitting MS The absence of other neurological, psychiatric or metabolic diseases besides MS.

Exclusion Criteria:

Exclusion criteria for this group included patients with exacerbation and/or steroid treatment in the last three months, as well as those with a history smoking, alcohol or sedative drug use, unstable vital signs, pregnancy, and serious health problems such as heart or kidney failure, major depression, severe anemia, immunodeficiency, narcolepsy, etc.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
Pure tone Audiometry Test | six month
  Air and bone conduction hearing thresholds will be measured using a Grason-Stadler GSI 61 Clinical Audiometer in a quiet room of the Industrial Acoustic Company (IAC) Inc. standard. Airway hearing thresholds will be measured using Telephonics TDH 39 headphones and bone conduction hearing thresholds will be measured using Radioear B-71 bone vibrator. Airway hearing thresholds will be evaluated at frequencies of 0.25 -8 kHz and bone conduction hearing thresholds at 0.5-4 kHz. As pure tone average, 500-1000-2000 Hz air and bone conduction thresholds will be calculated separately for both ears. A pure tone average between 0-15 dB will be considered normal hearing.
Speech Audiometry | six month
  Speech Audiometry will be performed in a quiet room to IAC (Industrial Acoustic Company) standards using a Grason-Stadler GSI 61 Clinical Audiometer.
  Speech reception threshold will be determined using three syllable word lists. A 40 dB Sensation Level (SL) will be added above the speech reception threshold and the patient will be asked if he/she can hear comfortably. After determining the level at which the patient can hear most comfortably, 25-word monosyllabic isophonic word lists will be read and the speech discrimination score will be calculated as a percentage. Individuals with a speech discrimination score of 88% and above and with an agreement between speech reception threshold and pure tone averages (SSO) will be included in the study.
Speech Discrimination in Noise Test | Six month
  The SDN test will be performed in a quiet room in accordance with the Industrial Acoustic Company (IAC) standard using the Grason-Stadler GSI 61 Clinical Audiometer. After pure tone audiometry and speech tests, the GKAE test will be performed. The speech in noise discrimination test will be performed with a signal-to-noise (S/N) ratio of +10 dB. A word list at 50 dB SL will be presented to the tested ear using live sound, while simultaneously white noise at 40 dB SL will be presented to the test ear (Beattie et al. 1997). This will be done for both ears. The speech in noise discrimination test scores will be calculated as percentages (%) for both ears.
Otoacoustic Emission Test | Six month
  TEOAE measurements of all individuals in the study and control groups will be performed using the computer-based Otodynamics ILO-V6 'cochlear emission analyzer' and software version 5.61 (Otodynamics, London). Adult TEOAE probe will be used for all OAE measurements. The probe will be calibrated in a 1 cc acoustic calibration cavity. The measurement will be performed by averaging the nonlinear, 80 µsec, 260 click stimulus response at 80 ± 3 dB SPL. "Noise rejection level of 47 dB, wave reproducibility of 70% or more, and stimulus stability greater than 80% will be taken into consideration.
Contralateral Suppression Test | Six month
  For TEOAE and contralateral suppression measurements, 60 dB SL white noise will be applied from the opposite ear using a TEOAE probe and emission amplitudes will be measured from the same side ear. All OAE measurements will be performed by inserting the probe once and TEOAE and contralateral suppression tests will be performed respectively. Amplitude (dB) values obtained with suppression at 1000, 1414, 2000, 2828 and 4000 Hz will be used as study parameters.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment Scale | Six Month
  Translated into Turkish as the Montreal Cognitive Assessment Scale and abbreviated as MOBID, MOCA assesses attention, executive/managerial functions, memory, visual-spatial skills, language, abstract thinking and arithmetic. It is easy and practical to apply. The score that can be obtained varies between 0-30. The cut-off point for cognitive impairment is 21. Patients who perform below 21 points are considered to have cognitive impairment. Although it is not a battery used in the MS patient group, a study conducted on 39 MS patients and 20 healthy people showed that it can be used safely for screening purposes in patients with MS (Aksoy et al., 2013; Nasreddine et al., 2005; Selekler & Cangoz, 2009).
Symbol Digit Modalities Test | Six Month
  Attention, visuospatial information processing speed and working memory are assessed. It is one of the subtests of the Short Repeatable Neuropsychological Battery developed to assess cognitive functions in MS (Smith, 1973).

CONTACTS AND LOCATIONS:
Overall Officials: ASUMAN KÜÇÜKÖNER, Dr., Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be published as a research article.